CLINICAL TRIAL: NCT04087382
Title: Mechanical Thrombectomy in Acute Ischemic Stroke Beyond the Time of Window: Non Randomized Controlled Clinical Trial
Brief Title: Mechanical Thrombectomy in Acute Ischemic Stroke Beyond the Time of Window
Acronym: AIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Collaborators: Ain Shams University (Other); Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Eman M. Khedr, Professor of Neurology, Assiut University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M thrombectomy in late AIS
Record Dates: First submitted 2019-09-06; First posted 2019-09-12 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Thrombectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): it included 32 patients with acute ischemic stroke beyond the time of window (more than 6 hours) assigned to mechanical thrombectomy) plus the conventional treatment (Aspirin 150 mg and atorvastatin 40 mg).
  Interventions: Device: thrombectomy
- non-intervention group (Other): it included 25 patients with acute ischemic stroke beyond the time of window (more than 6 hours) who received medical treatment (Aspirin 150 mg and atorvastatin 40 mg).
  Interventions: Other: non intervention group

INTERVENTIONS:
Device: thrombectomy — Transfemoral a microcatheter with its distal end was positioned a few millimeters beyond the distal aspect of the clot, the guide wire was exchanged by Solitaire stent device. The device was held in place when 3 mm was out of the microcatheter. The microcatheter was slowly pulled back to deploy the TR or ST device over the clot.
  Arms: Intervention group
Other: non intervention group — medical treatment (Asprin, statin, nootropic drug)
  Arms: non-intervention group

SUMMARY:
Background: intravenous alteplase appears to be much less effective at opening proximal occlusions of the major intracranial arteries, which account for more than one third of cases of acute anterior-circulation stroke and expanding time window using mechanical thrombectomy can improve clinical outcome in patients that would have only received conservative treatment.

The aim of this work is to evaluate the effectiveness of endovascular therapy within 24 hours of symptom onset and to compare clinical outcome of endovascular therapy with the standard medical therapy at the end of 3rd month follow up.

Material and Methods 57 subjects presenting with an acute ischemic stroke caused by occlusion of the proximal middle cerebral artery (M1 segment) or Internal carotid artery ( ICA segment) within 24 hours from symptom onset as documented by Ct, and or MRI perfusion were recruited consecutively from 2 University hospitals Ain shams University Hospital (32 Patients) and Aswan University (25 patients). Assessment of each subject was performed using NIHSS, and MRS, Aspect score, before intervention. Follow up was done using the same clinical scale one week and the 3 month after the onset.

Primary outcome NIHSS and MRS at the end of 3 month after the onset. secondary outcome complications (cerebral Hge) and death at 3 months.

DETAILED DESCRIPTION:
Background Expanding time window using the emerging technologies for mechanical thrombectomy can improve chances of achieving successful thrombectomy and improve clinical outcome in patients that would have only received conservative treatment. The aim of this work is to evaluate the effectiveness and safety of endovascular therapy within 24 hours of symptom onset and to compare clinical outcome of endovascular therapy and standard medical therapy at the end of 3rd month.

Subjects and Methods:

This is a multicenteric case-control clinical trial (Ain shams and Aswan university hospitals), comparing clinical improvement and mortality/morbidity in patients presenting with acute ischemic stroke stroke caused by occlusion of the proximal middle cerebral artery (M1 segment) or Internal carotid artery (distal ICA segment) within 24 hours from symptom onset.

Onset of stroke was defined as time they were last known to be well. Ischemic stroke is characterized by the sudden loss of blood circulation to an area of the brain, resulting in a corresponding loss of neurologic function. It included 57 patients with acute ischemic stroke due to large vessel occlusion (LVO) admitted either to neurology department of Ain shams university hospitals or Aswan university hospitals between during the period from Jan 2019 and August 2019

All patients were subjected to the following:

A) Clinical assessment:

Full history taking with special emphasis upon: Age and Sex of the patient, onset of symptoms; onset is defined as the point in time the patient was last seen well, presence of vascular risk factors, namely: diabetes mellitus, hypertension, cardiac diseases, dyslipidemia and smoking. History of receiving drugs prior to arrival to the hospital, especially anti-coagulants, and anti-platelets & IV thrombolytics.

Complete general and neurological assessment including: complete general examination including blood pressure measurement using mercurial sphygmomanometer and random blood sugar assessment, neurological examination on admission with NIHSS assessment to determine initial NIHSS, neurological deficit was measured using (NIHSS) obtained on discharge and on day 90 with the modified Rankin Scale (mRS) measured on discharge and after 3 months (Bonita and Beaglehole, 1988). A standard 12-lead ECG to delineate presence of ischemic changes or arrhythmias was also done Routine ER laboratory investigations including: complete blood count and coagulation profile and serum urea and creatinine.

Hypertension was defined as self-report of hypertension with antihypertensive medication use, and/or systolic blood pressure greater than or equal to 140 mm Hg, and/or diastolic blood pressure greater than or equal to 90 mm Hg. Diabetes was defined as being on treatment for diabetes by self-report with antidiabetic drugs and/or having a fasting glucose level greater than or equal to 126 mg/dL, plasma glucose ≥ 200 mg/dl 2 h after a 75-g oral glucose load as in a glucose tolerance test, or glycated hemoglobin (HbA1C) ≥ 6.5%. Patients with past or current history of smoking were categorized as smokers. Dyslipidemia was defined as serum total cholesterol (TC) > 240, serum LDL-c > 160, serum triglycerides (TAG) > 200 and/or serum HDL-c < 40 (WHO 2006).

B) Radiological assessment:

Early ischemic changes and collateral circulation were assessed with the Alberta stroke program for early computed tomography (CT) ischemic score (ASPECTS) and with computed tomography angiography (CTA), magnetic resonance angiography (MRA) or digital subtraction angiography (DSA) for localization of the LVO.

N.B: a CT scan was routinely performed between 24 and 36 h after treatment or before in case of any neurological worsening (≥4-point increase in NIHSS score) occurred.

Procedure of endovascular intervention:

All patients in the 1st group (vascular intervention group) underwent primary thrombectomy with either the Trevo (TR) stent or the Solitaire (ST) stent (according to the availability) within the first 24 hours of symptoms onset.

All procedures were performed under the investigator's institutional mild sedation protocol. Some cases needed general anesthesia.

Favorable outcome was defined as achieving functional independence "mRS of 0,1or 2 in 3 months, poor outcome was defined as mRS of 3-5. Treatment starting is defined as femoral puncture.

Vascular recanalization was defined as thrombolysis in cerebral ischemia (TICI) score. Successful recanalization was defined as TICI grade 2b to 3.

Established device-related complications, namely, vascular perforation, arterial dissection, or embolization, were systematically collected. Symptomatic intracranial hemorrhage was defined as a hemorrhagic transformation on the 24-h computed tomography (CT) scan related to the deterioration in the patient's clinical condition in the judgment of the clinical investigator.Statistical analysis:

Statistical analysis was performed using the Statistical Package for the Social Sciences (IBM SPSS statistics V23).

Adjusted for age group (1=<70, 2= ≤70 years), Sex (female=0 or male=1), Diabetes mellitus (yes=1 or no=0), Hypertension (yes=1 or no=0),Cardiac (AF=1, IHD=2, Rheumatic heart=3, normal =4, AF +IHD =5) Smoking (yes=1 or no=0), Dyslipidemia (yes=1 or no=0), (B, correlation coefficient; CI, confidence interval; OR, odds ratio; SE, standard error; Wald statistics for logistic regression analysis.

The outcome of interest was the change in NIHSS and mRS scores throughout 90 days. Continuous variables are expressed as mean + standard deviation and categorical variables with percentage of occurrence. For comparison of continuous variables, the Mann-Whitney test was used between-group comparison. Chi Square test was used for analysis of proportions. A p Value <0.05 was the threshold for statistical significance.

ELIGIBILITY:
Inclusion criteria

1. Patients Aged between 18 and 80 years old.
2. Patients with acute ischemic stroke due to occlusion of the MCA or ICA suitable for endovascular treatment, as evidenced by CTA, MRA or angiogram.

4. Patients with symptoms onset between 6- 24 hours from arrival to the time of femoral puncture.

Exclusion criteria

A. Clinical exclusion criteria:

1. Patients known to have hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with INR > 2.0.
2. Patients with a pre-existing neurological or psychiatric disease that would confound the neurological evaluations; mRS score before the onset of stroke must be ≤ 1.

B. Neuroimaging exclusion criteria:

1. Patients with hypodensity on CT accounting to an ASPECTS score of <7.
2. Patients with CT or MRI evidence of hemorrhage (the presence of micro-bleeds is allowed).
3. Patients Significant mass effect with midline shift on CT brain.
4. Subjects with occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior/posterior circulation) on CT brain.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
1- Measuring the Modified Rankin Score (MRS) on day 90 | 3 months
  1- Measuring the Modified Rankin Score (MRS) on day 90 (ranging from, 0 to 6, with higher scores indicating greater disability). Favorable outcome was defined as achieving functional independence (mRS of 0,1or 2) poor outcome was defined as MRS of 3-5.
2- Measuring the changes in NIHSS on day 90 | 3 months
  2- Changes in National Institute of Health Stroke Scale (NIHSS) were also measured at baseline (pre-thrombectomy) and on day 90. Favorable outcome when the score decrease by 4 or more point of the score.

SECONDARY OUTCOMES:
1-Estimate the number and percent of participants who have vascular recanalization | 3 months
  1-Estimate the number and percent of patients who have vascular recanalization according to thrombolysis in cerebral ischemia (TICI) score. TICI categories span from no perfusion (grade 0) to complete perfusion (grade 3). The "partial perfusion" category (grade 2) is defined as cases in which contrast passes the obstruction but with rates of entry and wash-out slower than normal and is subdivided into 2 subcategories, 2a and 2b. Successful vascular recanalization was defined as TICI grade 2b to 3.
2- Estimate the number of participants who developed complications | 3 months
  2-estimate the number of patients who developed complication death (mRS=6) symptomatic intracerebral hemorrhage, and arterial dissection.

CONTACTS AND LOCATIONS:
Overall Officials: Eman M khedr, Professor, Principal Investigator — Assiut University
Locations (2):
- Egypt (2):
  - Ahmed El-Bassiony, Cairo, Cairo, Egypt
  - Abdalla Khalil, Aswān, Select State/Province

REFERENCES:
- [Background] Albers GW, Marks MP, Kemp S, Christensen S, Tsai JP, Ortega-Gutierrez S, McTaggart RA, Torbey MT, Kim-Tenser M, Leslie-Mazwi T, Sarraj A, Kasner SE, Ansari SA, Yeatts SD, Hamilton S, Mlynash M, Heit JJ, Zaharchuk G, Kim S, Carrozzella J, Palesch YY, Demchuk AM, Bammer R, Lavori PW, Broderick JP, Lansberg MG; DEFUSE 3 Investigators. Thrombectomy for Stroke at 6 to 16 Hours with Selection by Perfusion Imaging. N Engl J Med. 2018 Feb 22;378(8):708-718. doi: 10.1056/NEJMoa1713973. Epub 2018 Jan 24. PMID 29364767
- [Background] Khedr EM, Fawi G, Abdela M, Mohammed TA, Ahmed MA, El-Fetoh NA, Zaki AF. Prevalence of ischemic and hemorrhagic strokes in Qena Governorate, Egypt: community-based study. J Stroke Cerebrovasc Dis. 2014 Aug;23(7):1843-8. doi: 10.1016/j.jstrokecerebrovasdis.2014.03.001. Epub 2014 Jun 21. PMID 24957312
- [Background] Vidale S, Longoni M, Valvassori L, Agostoni E. Mechanical Thrombectomy in Strokes with Large-Vessel Occlusion Beyond 6 Hours: A Pooled Analysis of Randomized Trials. J Clin Neurol. 2018 Jul;14(3):407-412. doi: 10.3988/jcn.2018.14.3.407. PMID 29971982
- [Background] Saver JL, Jahan R, Levy EI, Jovin TG, Baxter B, Nogueira RG, Clark W, Budzik R, Zaidat OO; SWIFT Trialists. Solitaire flow restoration device versus the Merci Retriever in patients with acute ischaemic stroke (SWIFT): a randomised, parallel-group, non-inferiority trial. Lancet. 2012 Oct 6;380(9849):1241-9. doi: 10.1016/S0140-6736(12)61384-1. Epub 2012 Aug 26. PMID 22932715
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL; American Heart Association Stroke Council. 2018 Guidelines for the Early Management of Patients With Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2018 Mar;49(3):e46-e110. doi: 10.1161/STR.0000000000000158. Epub 2018 Jan 24. PMID 29367334
- [Background] Smith EE, Saver JL, Cox M, Liang L, Matsouaka R, Xian Y, Bhatt DL, Fonarow GC, Schwamm LH. Increase in Endovascular Therapy in Get With The Guidelines-Stroke After the Publication of Pivotal Trials. Circulation. 2017 Dec 12;136(24):2303-2310. doi: 10.1161/CIRCULATIONAHA.117.031097. Epub 2017 Oct 5. PMID 28982689
- [Background] Saver JL, Goyal M, van der Lugt A, Menon BK, Majoie CB, Dippel DW, Campbell BC, Nogueira RG, Demchuk AM, Tomasello A, Cardona P, Devlin TG, Frei DF, du Mesnil de Rochemont R, Berkhemer OA, Jovin TG, Siddiqui AH, van Zwam WH, Davis SM, Castano C, Sapkota BL, Fransen PS, Molina C, van Oostenbrugge RJ, Chamorro A, Lingsma H, Silver FL, Donnan GA, Shuaib A, Brown S, Stouch B, Mitchell PJ, Davalos A, Roos YB, Hill MD; HERMES Collaborators. Time to Treatment With Endovascular Thrombectomy and Outcomes From Ischemic Stroke: A Meta-analysis. JAMA. 2016 Sep 27;316(12):1279-88. doi: 10.1001/jama.2016.13647. PMID 27673305
- [Background] Goyal M, Menon BK, van Zwam WH, Dippel DW, Mitchell PJ, Demchuk AM, Davalos A, Majoie CB, van der Lugt A, de Miquel MA, Donnan GA, Roos YB, Bonafe A, Jahan R, Diener HC, van den Berg LA, Levy EI, Berkhemer OA, Pereira VM, Rempel J, Millan M, Davis SM, Roy D, Thornton J, Roman LS, Ribo M, Beumer D, Stouch B, Brown S, Campbell BC, van Oostenbrugge RJ, Saver JL, Hill MD, Jovin TG; HERMES collaborators. Endovascular thrombectomy after large-vessel ischaemic stroke: a meta-analysis of individual patient data from five randomised trials. Lancet. 2016 Apr 23;387(10029):1723-31. doi: 10.1016/S0140-6736(16)00163-X. Epub 2016 Feb 18. PMID 26898852